CLINICAL TRIAL: NCT07090018
Title: A Pilot Feasibility Trial for an Intervention to Reduce Chronic Pain Following Cesarean Delivery
Brief Title: Empowered Relief: A One-Time Session to Help Postpartum Women Manage Ongoing Pain After Cesarean Delivery
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Principal Investigator, PSultan, Professor of Anesthesiology, Perioperative and Pain Medicine (Obstetrics), Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 80475; 1R90HD118650 (NIH)
Record Dates: First submitted 2025-07-22; First posted 2025-07-29 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-07

CONDITIONS: Chronic Pain; Cesarean Section Complications
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1-Session pain relief skills session (Empowered Relief) (Experimental): Participants will attend an Empowered Relief session at the beginning of the study period.
  Empowered Relief is a 2-hour one session pain relief skills intervention that is delivered to patients by a certified instructor using a standardized treatment manual and slide deck. Content includes completion of a pain survey, pain neuroscience education, information on pain and stress responses, experiential exercises, information on three core pain management skills, completion of a personalized plan for empowered relief, and receipt of a binaural app for daily use.
  Standard of care will be maintained for all participants, and supplemented with Empowered Relief. Pain management is not a factor for inclusion/exclusion criteria and patients will continue their pain management as prescribed and directed by their provider
  Interventions: Behavioral: Empowered Relief
- Control arm: Postpartum Standard of Care (No Intervention): Participants will follow their current standard of care.

INTERVENTIONS:
Behavioral: Empowered Relief — The participants will attend a pain relief skills intervention (Empowered Relief). The two-hour session is delivered by a certified instructor and includes pain neuroscience education, 3 core pain management skills, experiential exercises, completion of a personalized plan for empowered relief. Participants download a binaural relaxation audio file for daily use.
  Other Names: 1-Session Pain Relief Skills Intervention
  Arms: 1-Session pain relief skills session (Empowered Relief)

SUMMARY:
The purpose of this study is to study the effect of a pain relief skills session (Empowered Relief) on chronic pain incidence at 12 weeks post cesarean delivery.

ELIGIBILITY:
Inclusion Criteria:

* Females 18 years of age or older
* Any postpartum woman who has had a cesarean delivery in the Stanford Healthcare system with a viable birth
* has moderate/severe pain, scoring ≥ 4/10 on the numerical/visual analog scale that continues at 6 weeks postpartum
* English fluency
* Ability to adhere to and complete study protocols
* Access to smart device for zoom / video meetings

Exclusion Criteria:

* <18yrs
* Chronic pain prior to pregnancy
* Cognitive impairment, non-English speaking, or psychological factors that would preclude comprehension of material and/or full participation in the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 60 (Estimated)
Dates: Start 2025-09-25 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of participants registering for Empowered Relief session | Baseline (up to 1 week)
Percentage of participants attending Empowered Relief session | Treatment (up to 2 weeks)
Participant Satisfaction Scale Score | 1 - 2 weeks Post treatment
  Participant satisfaction will be measured using a 7 item questionnaire (scale ranges from 0 - 42, higher ratings represent greater satisfaction with the treatment).
Participant Treatment Skills Use Scale Score | 4 - 6 weeks Post Treatment
  Participant treatment skills use will be measured with a 5 items questionnaire (scale ranges from 0 - 25, higher ratings represent increased time using treatment).

SECONDARY OUTCOMES:
Change from baseline in PROMIS Pain Interference 8a scale score | Baseline, Week 6
  Participants complete Patient Reported Outcomes Measurement Outcomes System (PROMIS) Pain Interference 8a questionnaire, an 8-item scale assessing pain interference with life enjoyment, concentration, and daily activities over the past 7 days.
  (Score range 8 - 40, higher scores represent a greater degree of pain interference).
Change from baseline in PROMIS Pain Intensity 3a scale score | Baseline, Week 6
  Participants complete PROMIS Pain Intensity 3a questionnaire, a 3-item scale assessing average pain intensity for the past 7 days.
  (Score range 3 - 15, higher score represents a greater degree of pain intensity)
Change from baseline in Pain Catastrophizing Scale Score | Baseline, Week 6
  Participants complete Pain Catastrophizing questionnaire, a 13-item scale assessing an individual's pain experience
  (Score range 0 - 52, higher score represents a greater degree of pain catastrophizing)
Change from baseline in PEG scale score (composite) | From enrollment to the end of study completion at 6 weeks
  Participants complete thrice weekly Pain, Enjoyment, General Activity Scale (PEG) questionnaire, a 3-item scale assessing pain interference and intensity via SMS.
  (Score range 0 - 30, higher score represents a greater degree of pain intensity/interference)
Change from baseline in PEG scale score (pain interference) | From enrollment to the end of study completion at 6 weeks
  Participants complete thrice weekly PEG questionnaire, to assess pain interference via SMS.
  (Score range 0 - 20, higher score represents a greater degree of interference)
Change from baseline in PEG scale score (pain intensity) | From enrollment to the end of study completion at 6 weeks
  Participants complete thrice weekly PEG questionnaire to assess pain intensity, via SMS.
  (Score range 0 - 10, higher score represents a greater degree of pain intensity)
Response rate to individual items of the PEG scale score via SMS | From enrollment to the end of study completion at 6 weeks
  Participant percentage responding to items of the thrice weekly PEG questionnaire, a 3-item scale assessing pain interference and intensity via SMS.
  (Score range 0 - 3; higher scores indicate higher response rate)

CONTACTS AND LOCATIONS:
Overall Officials: Pervez Sultan, MBChB, FRCA, MD(Res), Principal Investigator — Stanford University
Locations (1):
- Stanford University, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol
Time Frame: Beginning 9 months and ending 36 months following article publication.
Access Criteria: Wish whom? Investigators whose proposed use of the data has been approved by an independent review committee ("learned intermediary") identified for this purpose.
  For what types of analysis? For individual participant data meta-analysis
  By what mechanism will data be made available? Proposals may be submitted up to 36 months following article publication. After 36 months the data will be available in our University's data warehouse but without investigator support other than deposited metadata. Information regarding submitting proposals and accessing data may be found at (Link to be provided).

REFERENCES:
- [Background] Ciechanowicz S, Joy RR, Kasmirski J, Blake L, Carvalho B, Sultan P. Incidence, Severity, and Interference of Chronic Postsurgical Pain After Cesarean Delivery: A Systematic Review and Meta-analysis. J Clin Anesth. 2025 Jun;104:111832. doi: 10.1016/j.jclinane.2025.111832. Epub 2025 Apr 24. PMID 40279839